CLINICAL TRIAL: NCT06327295
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the
Brief Title: A Study of ATB1651 in Adults With Mild to Moderate Onchomycosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AmtixBio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATB1651-102
Record Dates: First submitted 2024-02-29; First posted 2024-03-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ATB1651-102 Cohort 1 (Experimental): The planned ATB1651 dose of 3% solution to each infected toenail once daily for 12 weeks (follow up for 24 weeks) Twenty-five participants are expected to enroll per cohort.
  Interventions: Drug: ATB1651-102- Cohort 1
- ATB1651-102 Cohort 2 (Experimental): The planned ATB1651 dose of 3% solution to each infected toenail once daily for 20 weeks follow up for 16 weeks) Twenty-five participants are expected to enroll per cohort.
  Interventions: Drug: ATB1651-102- Cohort 2
- ATB1651-102 Cohort 3 (Experimental): The planned ATB1651 dose of 3% solution to each infected toenail twice daily for 12weeks follow up for 24 weeks).
  Twenty-five participants are expected to enroll per cohort.
  Interventions: Drug: ATB1651-102- Cohort 3
- ATB1651-102 Cohort 4 (Experimental): The planned ATB1651 dose of 5% solution to each infected toenail once daily for 12weeks follow up for 24 weeks).
  Twenty-five participants are expected to enroll per cohort.
  Interventions: Drug: ATB1651-102- Cohort 4
- Placebo (Placebo Comparator): Matching placebo to the IP per cohort.
  Five participants are expected to be enrolled per cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATB1651-102- Cohort 1 — Dosage form- Topical solution; Dosage- 3% formulation The participants will apply the daily dose of 3% ATB1651 once daily to the affected great toenail for 12 weeks with a follow-up for 24 weeks.
  Arms: ATB1651-102 Cohort 1
Drug: ATB1651-102- Cohort 2 — Dosage form- Topical solution; Dosage- 3% formulation The participants will apply the daily dose of 3% ATB1651 once daily to the affected great toenail for 20 weeks with a follow-up for 16 weeks.
  Arms: ATB1651-102 Cohort 2
Drug: ATB1651-102- Cohort 3 — Dosage form- Topical solution; Dosage- 3% formulation The participants will apply the daily dose of 3% ATB1651 twice daily to the affected great toenail for 12 weeks with a follow-up for 24 weeks.
  Arms: ATB1651-102 Cohort 3
Drug: ATB1651-102- Cohort 4 — Dosage form- Topical solution; Dosage- 5% formulation The participants will apply the daily dose of 5% ATB1651 once daily to the affected great toenail for 12 weeks with a follow-up for 24 weeks.
  Arms: ATB1651-102 Cohort 4
Drug: Placebo — participants will receive matching placebo across cohorts 1-4 of the study.
  Arms: Placebo

SUMMARY:
The study is designed to evaluate the Safety, Tolerability and Pharmacokinetics of ATB1651 in participants with mild to moderate onychomycosis

DETAILED DESCRIPTION:
This Phase 2, multicenter, randomized, double-blind, placebo-controlled study is designed to assess the efficacy, safety, and tolerability of ATB1651 when administered topically to the great (hallux) toenail of participants with mild to moderate onychomycosis who are otherwise healthy.

This study will enroll upto 120 participants in 3+1 (optional) sequential cohorts.

* Participants in Cohorts 1 to 3 will be randomized within each cohort to receive either ATB1651 3% or placebo at a ratio of 5:1.
* An optional cohort (Cohort 4) may enroll up to 30 participants who will be randomized to receive either ATB1651 5% or placebo at a ratio of 5:1.

Dosing will start with Cohort 1 followed at least 4 weeks later by Cohort 2. The decision to continue dosing in Cohort 2 beyond 12 weeks and/or to commence Cohort 3, at the planned dosage regimen or a modified dosage regimen, will be determined by the Safety Review Committee (SRC).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of onychomycosis by positive mycological (KOH) staining and positive culture from affected great toenail(s).
2. Appearance of onychomycosis involving 20% to 60% of 1 (or both) affected great toenail(s), as determined by visual inspection after the nail has been trimmed. If the percentage of infection is outside this range but is still considered appropriate for this study, based on the overall impression of the Principal Investigator (PI), participation can be considered in consultation with the Medical Monitor (MM). The visual inspection results of the appearance of onychomycosis involving 20% to 60% of 1 (or both) affected great toenail(s) will be reviewed by the Sponsor before enrollment.
3. The combined thickness of the distal nail plate at the associated hyperkeratotic nail bed is < 2 mm.
4. Adult males and females, 18 to 70 years of age (inclusive) at the time of Screening.
5. In good general health, with no significant medical history, and no clinically significant abnormalities on physical examination or ECG at Screening and/or before the first administration of IP at the discretion of the PI or designee. Participants with mild stable disease may be considered eligible at the discretion of the PI or designee.
6. Body mass index (BMI) between 17.5 and 35.0 kg/m2, inclusive, at Screening.

Exclusion Criteria:

1. History of allergy to any of the excipients in ATB1651.
2. Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at Screening or Day 1.
3. Underlying physical or psychological medical conditions that, in the opinion of the PI, would make it unlikely for the participant to comply with the protocol or complete the study per protocol.
4. Unwilling to refrain from the use of nail cosmetics such as clear and/ or colored nail lacquers from the Screening visit until the end of the study.
5. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half-lives of the product (whichever is the longest) or participation in more than 4 investigational drug studies within 1 year prior to Screening.
6. Diabetes mellitus requiring treatment other than diet and exercise.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the complete cure rate with topical ATB1651 3% and ATB1651 5% in participants with mild to moderate onychomycosis. | From screening to end of study treatment up to 252 days
  Complete cure rate (defined as 100% clear nail surface area for the target toenail at Week 36 and negative mycological evaluation of the affected great toe after the last dosing).

SECONDARY OUTCOMES:
To further evaluate the efficacy of topical ATB1651 3% and topical ATB1651 5% in participants with mild to moderate onychomycosis. | From screening to end of study treatment up to 252 days
  Efficacy of ATB1651 assessed based on Mycological evaluation of the affected great toenail(s) where ATB1651 was applied.
  Standardized high-resolution photographs will also be taken and provided to a central reader to confirm the measurements Fungal growth will be measured for the affected great toenail(s) by direct mycological examination using staining (KOH) and culture of the nail scrapings for Trichophyton rubrum, Trichophyton mentagrophytes, Candida albicans, and other fungal species.
To assess and collect the percentage and severity of adverse events (AEs). | From screening to end of study treatment up to 252 days
  Adverse Events include changes pain, erythema and local irritation, and clinically significant results from physical examinations. AE will be coded using the most current version of Medical Dictionary for Regulatory Activities (MedDRA®) Version 22.0 or higher.
Maximum plasma concentration (Cmax) | Cohort 1, 3 and 4- On day1, day 14, day 28, day 42, Day 56, day 70 and day 84; Cohort 2- Same as cohort 1+day 98, 112, day 126 and day 140
  Pharmacokinetic profile characterized by systemic exposure following multiple doses of ATB1651 by CMAX of ATB1651
Time to maximum plasma concentration (Tmax) | Cohort 1, 3 and 4- On day1, day 14, day 28, day 42, Day 56, day 70 and day 84; Cohort 2- Same as cohort 1+day 98, 112, day 126 and day 140
  Pharmacokinetic profile characterized by systemic exposure following multiple doses of ATB1651 through Tmax of ATB1651
Apparent terminal elimination rate constant (λz) | Cohort 1, 3 and 4- On day1, day 14, day 28, day 42, Day 56, day 70 and day 84; Cohort 2- Same as cohort 1+day 98, 112, day 126 and day 140
  Pharmacokinetic profile characterized by systemic exposure following multiple doses of ATB1651 by Apparent terminal elimination rate constant (λz)
Area under curve (AUC) | Cohort 1, 3 and 4- On day1, day 14, day 28, day 42, Day 56, day 70 and day 84; Cohort 2- Same as cohort 1+day 98, 112, day 126 and day 140
  Pharmacokinetic profile characterized by systemic exposure following multiple doses of ATB1651 by AUC
Apparent terminal half-life (t 1/2) | Cohort 1, 3 and 5- On day1, day 14, day 28, day 42, Day 56, day 70 and day 84; Cohort 2- Same as cohort 1+day 98, 112, day 126 and day 140
  Pharmacokinetic profile characterized by systemic exposure following multiple doses of ATB1651 by (t 1/2)
Apparent clearance (CL) | Cohort 1, 3 and 4- On day1, day 14, day 28, day 42, Day 56, day 70 and day 84; Cohort 2- Same as cohort 1+day 98, 112, day 126 and day 140
  Pharmacokinetic profile characterized by systemic exposure following multiple doses of ATB1651 by apparent clearance (CL).
Apparent terminal volume of distribution (VD) | Cohort 1, 3 and 4- On day1, day 14, day 28, day 42, Day 56, day 70 and day 84; Cohort 2- Same as cohort 1+day 98, 112, day 126 and day 140
  Pharmacokinetic profile characterized by systemic exposure following multiple doses of ATB1651 by VD
Plasma ATB1651 trough concentrations (Ctrough) | Cohort 1, 3 and 4- On day1, day 14, day 28, day 42, Day 56, day 70 and day 84; Cohort 2- Same as cohort 1+day 98, 112, day 126 and day 140
  Pharmacokinetic profile characterized by trough concentrations (Ctrough) of ATB1651

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research Christchurch, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No